CLINICAL TRIAL: NCT02508740
Title: Phase 1, Non-Randomized, Parallel-Group, Open-Label Study to Characterize the Pharmacokinetics of a Single Oral Dose of Bevenopran in Patients With Varying Degrees of Renal Impairment Compared to Healthy Subjects
Brief Title: Single Oral Dose of Bevenopran in Patients With Varying Degrees of Renal Impairment
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Development of compound has been put on hold.
Sponsor: Cubist Pharmaceuticals LLC, a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA) (Industry)
Collaborators: Syneos Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 5945-REN-13-03
Record Dates: First submitted 2015-07-22; First posted 2015-07-27 (Estimated); Last update posted 2015-07-27 (Estimated); Status verified 2015-07

CONDITIONS: Renal Impairment
MeSH Terms: conditions — Renal Insufficiency | interventions — DAC 5945

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- normal renal function (Experimental): Healthy subjects with normal renal function (Stage 1, >90 mL/min) will receive a single oral dose of 0.25 mg bevenopran.
  Interventions: Drug: bevenopran
- mild renal impairment (Experimental): Patients with mild renal impairment (Stage 2, 60-89 mL/min) will receive a single oral dose of 0.25 mg bevenopran.
  Interventions: Drug: bevenopran
- moderate renal impairment (Experimental): Patients with moderate renal impairment (Stage 3, 30-59 mL/min) will receive a single oral dose of 0.25 mg bevenopran.
  Interventions: Drug: bevenopran
- severe renal impairment (Experimental): Patients with severe renal impairment (Stage 4, <30 mL/min) will receive a single oral dose of 0.25 mg bevenopran.
  Interventions: Drug: bevenopran
- End Stage Renal Disease (ESRD) (Experimental): Patients with End Stage Renal Disease (ESRD) receiving dialysis for at least 3 months preceding the initial dose in this study (Stage 5) will participate in 2 treatment periods and will receive a single oral dose of 0.25 mg bevenopran at 3 hours after completion of the last hemodialysis session of the week in Period 1 and a single oral dose of 0.25 mg bevenopran at 3 hours before initiation of the last hemodialysis session of the week in Period 2
  Interventions: Drug: bevenopran

INTERVENTIONS:
Drug: bevenopran — Single oral dose
  Other Names: 5945

SUMMARY:
The purpose of this study is to characterize the effect of renal function on the PK of a 0.25 mg single oral dose of bevenopran in humans and to assess the safety and tolerability of bevenopran in patients with varying degrees of renal impairment and in healthy subjects.

DETAILED DESCRIPTION:
The current Food and Drug Administration (FDA) draft guidance for renal impairment studies advises performance of a PK study in patients with renal impairment for medications primarily excreted in urine and also for medications primarily metabolized or secreted in bile. The major routes of excretion of bevenopran in animals were identified as hepatobiliary and renal. In addition, preliminary findings show >40% of an oral bevenopran dose is eliminated unchanged in urine over a 48-72 hour period post-dose.

This is a Phase 1, non-randomized, parallel group, open-label study to characterize the effect of renal function on the PK of bevenopran in 1 or more study centers. At screening, eligible subjects will be enrolled and assigned to 1 of 5 parallel study groups of approximately 8 to 12 subjects each based on the classification of the renal function using estimated glomerular filtration rate (eGFR) from the Modification of Diet in Renal Disease (MDRD) Study, as presented in the FDA guidance on renal impairment studies. There are 5 study groups based on eGFRs.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy (other than renal impairment) male or female subjects 18 to 80 years of age, inclusive;
2. Body mass index (BMI) within the range of 18.0 to 45.0 kg/m2, inclusive, and a minimum weight of at least 50.0 kg at Screening;
3. Patients with renal impairment are to have mild, moderate, or severe renal impairment, or ESRD patients requiring dialysis. ESRD patients requiring dialysis should have been receiving dialysis on a 3 times/week schedule for at least 3 months preceding the initial dose in this study;
4. For healthy subjects and non-dialysis patients: If female, subject is not pregnant (as confirmed by pregnancy test at Screening and Day -1) and not planning to become pregnant within 30 days of last study drug administration, non-lactating, and is either:

   1. Not of child bearing potential, defined as postmenopausal for at least one year or <60 years old with no menses for >1 year confirmed by follicle stimulating hormone (FSH), or surgically sterile due to bilateral tubal ligation, bilateral oophorectomy, or hysterectomy;
   2. Of childbearing potential and utilizes one of the following: abstinence, hormonal contraceptives from at least 3 months prior to Screening, intrauterine device (IUD), double barrier method (acceptable double barrier methods are male condom plus sponge/diaphragm/hormones/IUD, condom plus spermicide is not acceptable), in combination with an additional method of contraception for their male partners. Subjects must be willing to practice these methods for the duration of the trial and for at least 30 days after last study drug administration. For dialysis patients (Group E): If female, must not be of child bearing potential, defined as postmenopausal for at least one year or <60 years old with no menses for >1 year confirmed by follicle stimulating hormone (FSH) or subject medical history, or surgically sterile (ie, bilateral tubal ligation, bilateral oophorectomy, or hysterectomy);
5. Male subjects with female sexual partners, must be using and willing to continue using medically acceptable forms of contraception (abstinence, vasectomy, or male condom for subjects plus an additional method of contraception for their female partners) from Screening and for at least 30 days after the last study drug administration;
6. Non-smoker for at least 1 year prior to Screening, as determined by self-reported history;
7. Able to speak, read, and understand English sufficiently to understand the nature of the study, to provide written informed consent, prior to the initiation of any protocol-specific procedures;
8. Must be willing and able to abide by all study requirements and restrictions;
9. Must be willing to abstain from the following foods from 1 week prior to first study drug administration until the end of the study: grapefruit, pomegranate, pomelo and star fruit juice/products, as well as foods containing poppy seeds, Seville oranges, and/or drinks or food containing quinine (ie, tonic water);
10. Must be willing to refrain from consuming more than 450 mg of caffeine per day (equivalent to approximately 2.5 cups of drip coffee);
11. Must be willing to refrain from strenuous physical activity for 48 hours prior to each study visit and during inpatient stays at the research site;
12. Must be willing to abstain from blood donation during the study and for 30 days after completion of study or early termination.

Exclusion Criteria:

1. For healthy subjects: history or presence of any clinically significant illness (e.g., cardiovascular, pulmonary, hepatic, renal, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurologic, oncologic, musculoskeletal, or psychiatric) or any other condition, including clinically significant anemia, which in the opinion of the investigator would jeopardize the safety of the subject or the validity of the study results; For renally impaired patients: as above, except renal insufficiency and other related stable medical conditions within the renally impaired subject population (eg, hypertension, diabetes, which should be stable for at least 3 months preceding the initial dose of study drug in this study) are allowed;
2. Clinically significant abnormalities on physical examination, medical history, 12-lead electrocardiogram (ECG), vital signs, or laboratory values, as judged by the investigator or designee. Subjects with renal impairment should have clinical laboratory values consistent with their disease and approved by the investigator;
3. QTcF > 480 ms for renally impaired patients and > 450 ms for healthy subjects;
4. Surgical or medical condition that may interfere with the absorption, distribution, metabolism, or excretion of the study drug, as judged by the investigator or designee;
5. Evidence of clinically significant hepatic (all subjects) or renal (healthy subjects only) impairment including alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 1.5 × upper limit of normal (ULN) or bilirubin > 1 × ULN;
6. Hemoglobin <9 g/dL, unless not considered clinically significant in the opinion of the investigator;
7. History of severe allergic reaction (including anaphylaxis) to any food, medication, or bee sting or previous status asthmaticus;
8. Patients with renal impairment who are not on a chronic stable drug regimen, defined as starting a new drug or changing dosage within 14 days prior to administration of study drug, except for drugs that manage the hemodialysis;
9. Patients with fluctuating or rapidly deteriorating renal function. Assessment of the stability of the patient's renal function will be determined by the investigator;
10. Patient has a functioning renal transplant (patient may be included in the study if he or she had a failed renal transplant and is not taking immunosuppressants);
11. Current self-reported drug or alcohol dependence (excluding caffeine), including subjects who have been in a drug rehabilitation program in the 6 months prior to Screening;
12. Use of any prescription drug, over the counter (OTC) medication or supplement, including p-gp inhibitors, within the 14 days (30 days for p-gp inducers) prior to dosing until study completion/early termination, unless therapeutic (renal patients) or approved by the medical monitor;
13. Use of any opioid therapy within 14 days or 5 half-lives of the specific opioid drug (whichever is longer) before the scheduled administration of study medication. Subjects using opioids to help manage their disease will need to wash out for 5 half-lives.
14. Positive drug screen upon presentation at Screening or upon Check-in at admission;
15. Positive breath alcohol test upon presentation at Screening or upon Check-in at admission;
16. History of allergy or hypersensitivity to bevenopran, or related drugs;
17. For healthy subjects: positive for Hepatitis B, Hepatitis C, or human immunodeficiency virus (HIV); For renally impaired patients: positive for Hepatitis B or HIV. Patients with Hepatitis C with acceptable liver function tests (as judged by the investigator or designee) may be included;
18. Donated or lost more than 450 mL of blood (one unit) in the 60 days preceding (first) study medication administration;
19. Has received an investigational product in a clinical trial within 30 days or 5 half-lives, whichever is longer, prior to first drug administration or is concurrently enrolled in any other type of medical research, judged not to be scientifically or medically compatible with this study; An employee of the sponsor or research site personnel directly affiliated with this study or their immediate family members defined as a spouse, parent, child or sibling, whether biological or legally adopted;

21. A subject who, in the opinion of the investigator or designee, is not considered to be suitable and is unlikely to comply with the study restrictions or study protocol for any reason.

Ages: 18 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2013-09; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Plasma concentrations of a 0.25 mg single oral dose of bevenopran | pre-dose, 0-8, 8-12, 12-24, 24-48, 48-72, 72-96, 96-120 h post-dose
  To characterize the effect of renal function on the PK of a 0.25 mg single oral dose of bevenopran in humans

SECONDARY OUTCOMES:
Number of adverse events for subjects enrolled | 6 days
  To assess the safety and tolerability of bevenopran in patients with varying degrees of renal impairment and in healthy subjects.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - DaVita Clinical Research: Denver Clinical Research Unit, Lakewood, Colorado
  - DaVita Clinical Research: Minneapolis Research Unit, Minneapolis, Minnesota